CLINICAL TRIAL: NCT05425329
Title: Safety and Efficacy of a Probiotic Supplement: Focus on Lessening Gastrointestinal Distress in Endurance Athletes
Brief Title: Safety and Efficacy of a Probiotic Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-FY2020-304
Record Dates: First submitted 2022-05-16; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Gastrointestinal Discomfort

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic treatment (Experimental): P. acidilatici, CECT 7483, L. plantarum CECT 7484, L. plantarum CECT7485 in a ration of 1:1:1 at a dose of 3b cfu/day.
  Interventions: Dietary Supplement: I3.1
- Placebo treatment (Placebo Comparator): Capsules indistinguishable from intervention containing maltodextrin.
  Interventions: Dietary Supplement: Placebo treatment

INTERVENTIONS:
Dietary Supplement: I3.1 — Capsule containing bacterial strains Lactobacillus plantarum (CECT7484 and CECT7485) and Pediococcus acidilactici (CECT7483) at a ratio of 1:1:1.
  Arms: Probiotic treatment
Dietary Supplement: Placebo treatment — Capsule containing maltodextrin.
  Arms: Placebo treatment

SUMMARY:
Exercise-induced gastrointestinal dysfunction is common amongst endurance athletes and is characterized by gastrointestinal permeability, also known as "leaky gut." Probiotics have been shown to improve gut permeability through the secretion of mucin, immunoglobulin A and improvement in stability of tight junctions between epithelial cells. This study will determine the efficacy of a probiotic containing the bacterial strains P. acidilatici, CECT 7483, L. plantarum CECT 7484, L. plantarum CECT7485) in altering markers of gut inflammation and dysfunction, and symptoms of gastrointestinal distress.

DETAILED DESCRIPTION:
This study is a randomized, placebo-controlled, double-blinded crossover study where trained runners that experience moderate gastrointestinal discomfort with exhaustive runs will be subjected to the probiotic intervention/placebo supplementation for one month with a one month washout period. The intervention consists of the probiotic strains Lactobacillus plantarum (CECT7484 and CECT7485) and Pediococcus acidilactici (CECT7483) at a ratio of 1:1:1 at a dose of 3b cfu/day. Probiotic/Placebo capsules will be taken once daily. Biological samples and symptom data collection will be collected at baseline and after one month of probiotic/placebo supplementation. Data are also collected after an in-house treadmill run after one month of supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Males, females between 18-50 years of age
* Healthy and injury free as determined by screening questions and medical history
* Distance runners as determined by physical activity questionnaire; run = 15 miles/week, run = 3 time or more/week
* VO2max level of = 40ml/kg/min for males or = 35ml/kg/min for females
* Agree to maintain normal diet and exercise routine throughout study
* Agrees to collect stool samples as needed
* Agree to complete questionnaires, records

Exclusion Criteria:

* Women who are pregnant or breastfeeding, or plan to become pregnant during course of the study will not be included as the effect of probiotic on pregnancy and lactation is not established.
* Subjects with a known allergy to the test material (active and placebo)
* Subjects taking NSAIDs, Metformin, probiotics, or supplements that might alter the gut microbiome;these will be assessed individually. (Multivitamin and protein supplementation are allowed)
* Subject that have abnormal test results during screening.
* Alcohol or drug abuse within past year (alcohol can impair gut barrier).
* History of GI surgery within past year as it would alter the gut microbiome (excluding appendectomy and herniorrhaphy).
* Severe heart, liver, kidney, neurological, oncological or psychiatric disease, or immunosuppressed subjects will be excluded.
* Coeliac disease, inflammatory bowel disease or acute pancreatitis (all 3 can impair gut barrier)
* Regular use of antacid medication (can significantly alter microbiota)
* Subject following a low FODMAP (fermentable oligo-, di-, mono-saccharides and polyols) diet will be excluded as this dietary pattern can alter the intestinal response to exercise in some people.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Effect of probiotic supplementation on intestinal fatty acid binding protein (iFABP) levels. | 4 weeks
  Determine concentration (pg/ml) of iFABP in serum
Effect of probiotic supplementation on lipopolysaccharide binding protein (LBP) levels | 4 weeks
  Determine concentration (ng/ml) of LBP in serum
Effect of probiotic supplementation on zonulin levels | 4 weeks
  Determine concentration (ng/ml) of zonulin in serum
Effect of probiotic supplementation on calprotectin levels | 4 weeks
  Determine concentration (ug/g) of calprotectin in feces.

CONTACTS AND LOCATIONS:
Overall Officials: Marie van der Merwe, PhD, Principal Investigator — University of Memphis
Locations (1):
- University of Memphis, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No